CLINICAL TRIAL: NCT05219630
Title: Change in Symptom and Quality of Life in COPD by Budesonide/Glycopyrronium/Formoterol Fumarate Pressurized Metered Dose Inhaler (BGF pMDI)
Acronym: EBISU
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00033
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD, PRO, BGF pMDI, CAT, RWD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is primarily aimed to investigate whether PROs can be improved after the initiation of BGF pMDI in real world clinical settings. While the study is 12-weeks in duration, the initial 4-week period will be used to assess immediate onset of benefits while the full study length will serve to demonstrate durability in response.

Study design:

This is a 12-week, multi-center, prospective observational study in which a total number of 107 patients will be enrolled. Adult outpatients with COPD without asthma history and who initiate on BGF pMDI as decided by the physicians in their routine clinical care will be consecutively invited for this study. Investigators (physicians) make screening their patients prior to the study entry and make informed consent explanation at their usual visit timing to the all eligible patients. After fulfilling eligibility criteria at study entry, the patients are enrolled in the study and the investigators will follow up the patients as in routine clinical practice and collect the data at baseline, at week 4 and week 12.

Data Source(s):

The study sites will be selected where BGF pMDI is used as a treatment option for COPD patients. Investigators participating in the study evaluate lung function (i.e., spirometry) for COPD patients in a daily practice

Statistical Analysis:

All data including patient characteristics at baseline will be summarized using appropriate descriptive statistics. Where applicable, changes from baseline at each timepoint will also be summarized using descriptive statistics. A comprehensive statistical analysis plan (SAP) including more details will be prepared prior to the database lock.

DETAILED DESCRIPTION:
This study is primarily aimed to investigate whether PROs can be improved after the initiation of BGF pMDI in real world clinical settings. While the study is 12 weeks in duration, the initial 4 weeks will be used to assess immediate onset of benefits while the full study length will serve to demonstrate durability in response. To help contextualize the study result, KRONOS data will be referred where applicable.

Study Design:

This is a 12-week, prospective, multi-center, observational study in which a total number of 107 patients will be enrolled. Adult outpatients with COPD without asthma history and who initiate on BGF pMDI as decided by physician in their routine clinical care will be consecutively invited for this study.

The day of the initiation of BGF pMDI treatment is called baseline, and the timing of fulfilling the eligibility criteria at baseline day is called the study entry.

Investigators (physicians) make screening their candidate patients who will be on the new prescription of BGF pMDI prior to the study entry and make explanation on informed consent at their usual visit timing. After fulfilling eligibility criteria at study entry, the patients are enrolled in the study and the investigators will follow up the patients as in routine clinical practice, and collect the data at baseline, at week 4 [Week 3 (Day 21) to Week 7 (Day 49)] and week 12 [Week 10 (Day 70) to Week 14 (Day 98)].

Data Source(s):

The study sites will be selected where BGF pMDI is used as a treatment option for COPD patients. Investigators participating in the study evaluate lung function (i.e., spirometry) for COPD patients in a daily practice

Statistical Analysis:

All data including patient characteristics at baseline will be summarized using appropriate descriptive statistics. Where applicable, changes from baseline at each timepoint will also be summarized using descriptive statistics. A comprehensive statistical analysis plan (SAP) including more details will be prepared prior to the database lock.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥40 years old at study entry
2. Patients diagnosed with COPD (based on post-bronchodilator forced expiratory volume 11/flow volume curve percent predicted forced (FEV1/FVC)<70% in the past and current or former smokers with a smoking history of ≥10 pack-years in the past)
3. Patients who is on the new prescription of BGF pMDI 320/18/9.6µg twice daily as per the physician's decision, at baseline
4. Patients with CAT≥10 at study entry
5. Patients who are capable to fill PROs physically and/or mentally as judged by investigators
6. Patients who provide written informed consent prior to the study entry

Exclusion Criteria:

1. Patients diagnosed as asthma by investigator's judgement at and/or before study entry
2. Patients who participated in any interventional clinical studies and/or any relevant studies (quality of life (QoL) and respiratory researches) during the 12 weeks before the study entry and/or during this study
3. Patients who used ICS+LABA+LAMA therapy including open triple and closed triple before the study entry
4. Patients with history of exacerbation during 4 weeks before the study entry
5. Patients with very severe comorbidities or status which would impact on QoL evaluation judged by investigators (e.g., heart failure, malignancy, receiving home oxygen therapy, pneumonia)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Around 15 sites across Japan will participate in the study. At each site, the investigators (physicians) will enroll adult patients without asthma history with COPD who initiates BGF pMDI as per the physicians' decision and during an outpatient visit at the in the clinics/hospitals.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Mean changes from baseline in the CAT scores (total score) over week 12 | 12 weeks
  CAT scores will be analysed using a linear model including timepoint (baseline, post-baseline). Mean of available CAT scores over week 4 to 12 will be used as post-baseline in this analysis. Based on the linear model, contrast will be used to estimate the mean changes from baseline over 12 weeks, its 2-sided 95% confidence interval and p-value.

SECONDARY OUTCOMES:
Mean changes from baseline in the SGRQ scores (total score) over week 12 | 12 weeks
  SGRQ scores will be analysed using a linear model including timepoint (baseline, post-baseline). Mean of available SGRQ scores over week 4 to 12 will be used as post-baseline in this analysis. Based on the linear model, contrast will be used to estimate the mean changes from baseline over 12 weeks, its 2-sided 95% confidence interval and p-value.
Mean changes from baseline in the SGRQ scores (total score) at week 4 and 12 | 12 weeks
  SGRQ scores will be analysed using mixed model for repeated measures (MMRM) including timepoint (baseline, week 4, week 12). For week 4 and 12 timepoints, available data closest to the target timepoint will be used in this analysis. This model account for within-patient correlation, i.e., the non-independence of repeated measures within a same patient. Unstructured covariance structure will be assumed for the within-subject covariance. Based on the MMRM, contrasts will be used to estimate the mean changes from baseline at week 4 and 12, their 2-sided 95% confidence interval and p-value.
To assess the achievement of MCID of SGRQ at 4 and 12 weeks from the initiation of BGF pMDI in COPD patients | 12 weeks
  The number and proportion of patients who achieved changes from baseline greater than or equal to MCID in SGRQ scores (i.e., changes from baseline in SGRQ scores ≥4) at each timepoint will be summarized. The exact 95% confidence interval for the single proportion will also be presented.

CONTACTS AND LOCATIONS:
Locations (17):
- Japan (17):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Seto, Aichi-ken
  - Research Site, Tōon, Ehime
  - Research Site, Kurume, Fukuoka
  - Research Site, Tsuchiura, Ibaraki
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Matsusaka, Mie-ken
  - Research Site, Kashihara, Nara
  - Research Site, Chūō, Tokyo
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kagoshima
  - Research Site, Miyazaki
  - Research Site, Osaka
  - Research Site, Ōita

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials/studies via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Muro S, Hozawa S, Sugiura H, Yoshida Y, Makita N, Kato Y, Hirai T, Nishida K, Kawayama T. Real-world effectiveness of budesonide/glycopyrronium/formoterol fumarate metered dose inhaler on symptoms and quality of life in patients with COPD: EBISU study. Respir Investig. 2025 Sep;63(5):726-733. doi: 10.1016/j.resinv.2025.05.007. Epub 2025 Jun 11. PMID 40513294
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00033&attachmentIdentifier=4a428dd5-2287-4287-88c9-7c3b5f6e5f13&fileName=Ver1.0_EBISU_Study_Synopsis_fix.pdf&versionIdentifier=